CLINICAL TRIAL: NCT01740583
Title: A Feasibility Study of the Mitralign Annuloplasty System for the Treatment of Chronic Functional Mitral Valve Regurgitation
Brief Title: Mitralign Percutaneous Annuloplasty System for Chronic Functional Mitral Valve Regurgitation
Acronym: ALIGN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mitralign, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLPR-007
Record Dates: First submitted 2012-11-30; First posted 2012-12-04 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Mitral Valve Regurgitation
Keywords: mitral valve, regurgitation, annuloplasty
MeSH Terms: conditions — Mitral Valve Insufficiency; Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- annuloplasty (Experimental): All patients will receive treatment with the Mitralign Percutaneous Annuloplasty System (MPAS).
  Interventions: Device: percutaneous annuloplasty

INTERVENTIONS:
Device: percutaneous annuloplasty — plication of the mitral valve annulus

SUMMARY:
The purpose of this study is to test the safety and device performance of the Mitralign system ("MPAS") to treat functional mitral valve regurgitation.

DETAILED DESCRIPTION:
The ALIGN study is a single arm, prospective study. The objective of the study is to investigate the safety and performance of a catheter-based plication device intended to reduce the circumference of the dilated mitral valve. The study will enroll up to 50 subjects from up to 5 sites (Paraguay, Columbia, Dominican Republic, Brazil, and India) who will be followed for 36 months post index procedure. Enrollment is defined at the time the study device is inserted into the body and patients will be followed at 30 days, and Months 6, 12, 24 and 36 post index procedure.

ELIGIBILITY:
Inclusion Criteria:

* NYHA II-IV
* Structurally normal mitral valve
* At least Grade 2 mitral regurgitation
* Left ventricular ejection fraction not less than 20% and not greater than 45%
* Left ventricular end diastolic diameter not less than 5.0 cm and not greater than 7.5 cm

Exclusion Criteria:

* Pregnant or lactating female
* Mitral stenosis
* Mod/severe aortic stenosis or regurgitation
* Mod/severe tricuspid stenosis or regurgitation
* Endocarditis
* Previous mitral valve repair or MV replacement
* Bioprosthetic or mechanical aortic valve
* Known unstable angina or MI within 30 days prior to procedure
* CVA within past 6 months
* Known contraindications to blood transfusion, contrast dye, DAPT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2012-11; Primary Completion 2017-01 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Events (MAE) | within 30 days post procedure
  MAE defined as occurrence of any of the following: Mitral valve-related surgery/intervention, myocardial infarction, cardiac tamponade, stroke, device and/or procedure-related death

SECONDARY OUTCOMES:
Echocardiographic Outcomes | at 6 months
  Freedom from an increase in ventricular diameter

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Ebner, M.D., Principal Investigator — Sanatorio Italiano (The Italian Hospital)
Locations (8):
- Colombia (2):
  - Clinica CardioVID, Medellín, Antioquia
  - Antonio Dager, MD, Valle Del Cauca, Cali
- France (2):
  - Bordeaux Heart University Hospital, Bordeaux-Pessac
  - Clinique Pasteur, Toulouse
- Sanatorio Italiano, Asunción, Paraguay
- Poland (3):
  - American Heart of Poland S.A., Bielsko-Biala
  - Centrum Medyczne HZP, Poznan
  - Instytutem Kardiologii, Warsaw